CLINICAL TRIAL: NCT05211609
Title: Prevalence of High Plasmatic 3-O-Methyldopa Level in a Specific Population of Patients With a Symptomatology Compatible With AADC Deficiency (Aromatic L-Amino Acid Decarboxylase)
Brief Title: Prevalence of High Plasmatic 3OMethyldopa Level in a Specific Population of Patients With a Symptomatology Compatible With AADC Deficiency
Acronym: DOPADEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7953 R21_0521
Record Dates: First submitted 2021-12-17; First posted 2022-01-27 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Aromatic L-Amino Acid Decarboxylase Deficiency
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasmatic 3-O-Methyldopa Level (Experimental): Prevalence of High Plasmatic 3-O-Methyldopa Level in a Specific Population of Patients With a Symptomatology Compatible With AADC Deficiency (Aromatic L-Amino Acid Decarboxylase)
  Interventions: Diagnostic Test: Plasmatic 3-O-Methyldopa dosage

INTERVENTIONS:
Diagnostic Test: Plasmatic 3-O-Methyldopa dosage — Plasmatic 3-O-Methyldopa dosage

SUMMARY:
O-MethyDopa (3-OMD) is a metabolite of the Dopaminergic pathway that accumulates in case of a default in the neurotransmitter biosynthesis due to a key enzyme deficiency: Aromatic L-Amino Acid Decarboxylase (AADC) deficiency. 3-OMD is a validated biomarker specific for this AADC enzyme defect.

The purpose of this study is to assess the prevalence of the elevation of 3-OMD in a predominantly pediatric targeted population with symptoms compatible with AADC deficiency; that will allow us to specify the indications for this screening test according to the clinical symptoms of the patients with the aim, ultimately, of optimizing the diagnosis of AADC deficiency.

DETAILED DESCRIPTION:
-O-MethyDopa (3-OMD) is a metabolite of the Dopaminergic pathway that accumulates in case of a default in the neurotransmitter biosynthesis due to a key enzyme deficiency: Aromatic L-Amino Acid Decarboxylase (AADC) deficiency. 3-OMD is a validated biomarker specific for this AADC enzyme defect. (Chen et al., 2014, Chien et al., 2016, Brennenstuhl et al., 2019).

To date, the prevalence of the elevation of 3-OMD has been studied in neonatal screening of healthy newborns and in patients with a previously proven AADC deficiency but not in a target population. (Chen et al., 2014, Chien et al., 2016, Brennenstuhl et al., 2019, Kubaski et al., 2021). The prevalence of elevated plasma 3-OMD, a biomarker of cerebral monoamine neurotransmitters deficiency, has never been evaluated in a targeted population.

The AADC enzyme is encoded by the DDC (Dopa-Decarboxylase) gene. Pathogenic bi-allelic variations of the DDC gene are responsible for a dysfunction of the AADC enzyme, leading to a decrease in the synthesis of biogenic amine neurotransmitters (Dopamine, Serotonin).

AADC deficiency is a rare recessive genetic disease, with less than 200 cases published in the literature. The clinical signs begin in childhood are varied, with a broad phenotypic spectrum, reflecting the deficiency in biogenic amine neurotransmitters: motor impairment, neurodevelopmental abnormalities (delay in acquisitions, cognitive disorders and / or disorders of social interactions), dysautonomia, epileptic seizures. However, there are no specific clinical symptoms and evoking this diagnosis is tricky (Pearson et al., 2020).

A confirmation of the diagnosis requires at least 2 positive tests among: (i) analysis of the profile of cerebrospinal fluid (CSF) neurotransmitters by lumbar puncture (ii) enzymatic study of AADC (iii) genetic study of the DDC gene (Wassenberg et al. al., 2017). The cerebrospinal fluid (CSF) analysis is an invasive examination and the enzymatic study is performed in only a few laboratories. Therefore, it is largely admitted that this pathology is underdiagnosed (Brun et al, 2010, Brennenstuhl et al, 2019, Hyland et al. 2019).

The purpose of this study is to assess the prevalence of the elevation of 3-OMD in a predominantly pediatric targeted population with symptoms compatible with AADC deficiency; that will allow investigators to specify the indications for this screening test according to the clinical symptoms of the patients with the aim, ultimately, of optimizing the diagnosis of AADC deficiency.

Targeted screening of the disease via the measuring of the level of 3-OMD would allow for :

* an early diagnosis
* an adequate and pertinent therapeutic strategy, while avoiding inappropriate treatment due to lack of diagnosis, which can go as far as targeted treatment by gene therapy
* genetic counseling to families since there is a 25% risk of recurrence

Although the level of 3-OMD is a validated and specific biomarker of AADC deficiency, the blood assay is performed in very few laboratories in Europe. This assay was recently developed in the Biochemistry laboratory of the Montpellier University Hospital (Pr Cristol, Dr Badiou).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a neurodevelopmental disorder and presenting one of the following criteria:

   * Motor development delay
   * Cerebral palsy
   * Hypotonia / hypertonia
   * Movement disorders: Oculogyric crises, dystonia, hypokinesia / bradykinesia
   * Catatonia
   * Dysautonomia: ptosis, excessive sweating, intermittent hypothermia, nasal congestion, fluctuating blood pressure
   * Epileptic encephalopathy
   * Autism spectrum disorder
2. Absence of cerebral structural abnormality on MRI apart from corpus callosum abnormality, white matter non-specific abnormality or cerebral atrophy
3. Collection of informed consent signed by both parents or legal guardians and by the child if possible or formed consent signed by adult
4. Patient benefiting from a social security scheme

exclusion criteria

1. Patient who had already have a neurotransmitter profiling or a measure of AADC enzymatic activity
2. Patient with a clearly defined anoxo-ischemic history
3. Patient with issues in blood collection

Ages: 0 Days to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
change of plasmatic 3-OMD level beyond 25% of reference value, by age group (0 - 30 days old, 31 - 365 days old, 1 - 10 years old, > 10 years old) | Day 0
  The prevalence of high 3-OMD level, with 95% confidence interval, will be estimated in the specific population with the frequency of patients with high plasmatic 3-OMD level, over 25% of normal levels defined by age. days old, 31 - 365 days old, 1 - 10 years old, > 10 years old)

SECONDARY OUTCOMES:
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Motor Development Delay | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Motor Development Delay Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Cerebral Palsy | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Cerebral Palsy Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Hypertonia/Hypotonia | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Hypertonia/Hypotonia Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients Movement Disorder | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients Movement Disorder Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Catatonia | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Catatonia Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Dysautonomia | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Dysautonomia Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Epileptic Encephalopathy | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Epileptic Encephalopathy Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Autism Spectrum Disorder | Day 0
  Comparison of the frequency of high 3-OMD LEVEL among the phenotype of symptomatology of the patients with Autism Spectrum Disorder Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.
Considering a potential diagnosis of AADC deficiency obtained in current patient care, available besides this study | Day 0
  Considering a potential diagnosis of AADC deficiency obtained in current patient care, available besides this study Prevalence of abnormal high 3-OMD level will be compared between the different phenotypic groups with Chi2 test. Each phenotypic group will be compared to the pool of the other groups. Odds ratio and 95% confidence interval will be presented.
  Prevalence of AADC deficiency will be estimated in the population for which the diagnosis of AADC deficiency, realized in current patient care, will be available in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Agathe ROUBERTIE, PH, Principal Investigator — a-roubertie@chu-montpellier.fr
Locations (2):
- France (2):
  - Angers University Hospital, Angers
  - Chu de Toulouse, Toulouse